CLINICAL TRIAL: NCT06231303
Title: Gut Microbiota Dysbiosis in Lupus Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: Hager Zanaty (Other)
Responsible Party: Sponsor-Investigator, Hager Zanaty, Assistant lecturer of nephrology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Gut microbiota in LN
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gut Microbiota Dysbiosis in Lupus Nepheritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extraction and PCR amplification Microbial community genomic DNA extraction from fecal samples will be done using extraction kit in accordance with the manufacturer's instructions. The DNA extract will be checked on a 1% agarose gel, and the DNA concentration and purity will be determined using the NanoDrop 2000 UV-vis spectrophotometer.
  The hyper-variable region V3-V4 of the bacterial 16S rRNA gene will be amplified with the primer pair 338F (ACTCCTACGGGAGGCAGCAG) and 806R (GGACTACHVGGGTATCTAAT) on a PCR thermocycler. PCR amplification of the 16S rRNA gene will performed as follows:
  Initial denaturation at 95 ℃ for 3 min. 27 cycles of denaturing at 95 ℃ for 30 s, annealing at 55 ℃ for 30 s, and extension at 72 ℃ for 45 s.
  Final extension step at 72 ℃ for 10 min and incubation at 10 ℃. The PCR product will then be used to quantify different bacterial species in stool samples of patients and controls using real time PCR.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with lupus nepheritis
  Interventions: Genetic: DNA extraction and PCR amplification
- Healthy persons of the same age
  Interventions: Genetic: DNA extraction and PCR amplification

INTERVENTIONS:
Genetic: DNA extraction and PCR amplification — Microbial community genomic DNA extraction from fecal samples will be done using extraction kit in accordance with the manufacturer's instructions. The DNA extract will be checked on a 1% agarose gel, and the DNA concentration and purity will be determined using the NanoDrop 2000 UV-vis spectrophotometer.
  The hyper-variable region V3-V4 of the bacterial 16S rRNA gene will be amplified with the primer pair 338F (ACTCCTACGGGAGGCAGCAG) and 806R (GGACTACHVGGGTATCTAAT) on a PCR thermocycler. PCR amplification of the 16S rRNA gene will performed as follows:
  Initial denaturation at 95 ℃ for 3 min. 27 cycles of denaturing at 95 ℃ for 30 s, annealing at 55 ℃ for 30 s, and extension at 72 ℃ for 45 s.
  Final extension step at 72 ℃ for 10 min and incubation at 10 ℃. The PCR product will then be used to quantify different bacterial species in stool samples of patients and controls using real time PCR.

SUMMARY:
Evaluate dysbiosis of some intestinal microbiota in adult patients with lupus nephritis compared to healthy controls.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is an autoimmune disease resulting in multi-organ inflammation with complex clinical manifestation including neuropsychiatric, lupus nephritis..etc. However, the actual cause of SLE is still unknown [1].

Various etiologies have been postulated which can be categorized into genetic and environmental such as age, gender, ultra-violet exposure, dietary intake, alcohol, and lifestyle behavior [2].

Lupus nephritis is one of the most severe manifestations of SLE with high mortality rate and 10% of them eventually develop end-stage renal disease within 5 years after diagnosis [3,4].

There are trillion of microbes inhabited human gut which dominated by 4 phyla; Firmicutes, Bacteroidetes, Proteobacteria and Actinobacteria. In healthy human gut, 98% of gut microbiota is dominated by Bacteroidetes and Firmicutes. Every species of gut microbiota play their own role in modulating immune system. Many factors could alter gut communities such as infant transition, dietary habit, age, gender and antibiotic consumption [5, 6].

Firmicutes responsive in fatty acids and carbohydrates absorption whereas Bacteroidetes correspond to polysaccharides absorption [7].

Recently, enormous reports highlighted on the association of autoimmune diseases with dysbiosis of gut microbiota [8-11], During the autoimmune disease condition, the symbiotic relationship is broken due to various factor such as dietary habit that change microbiota diversity. The decrease of microbial diversity was found in autoimmune diseases such as SLE and inflammatory bowel disease (IBD), presented by reduce commensal bacteria (Firmicutes and Bacteroidetes) and increase of detrimental bacteria (Proteobacteria and Actinobacteria) [12].

Alteration of gut microbiota expresses as Firmicutes/Bacteroidetes ratio (F/B) potentially act as the measurement for pathological condition in SLE patients which cause systemic inflammation. The decreased ratio of F/B microbiome in SLE patients occur either by the reduction in Firmicutes or increase abundance of Bacteroidetes [13]. In human study, altered short chain fatty acids (SCFA) fecal level in lupus patient with low F/B ratio suggest the potential link of gut absorption function with microbes [14].

Hence, it is necessary to identify the exact mechanism on how the gut microbiota promote SLE and LN pathogenesis in human studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients diagnosed with lupus nephritis. Adult age and sex matched healthy individuals will be included as a control group.

Informed consent will be obtained from each study participant.

Exclusion Criteria:

* Subjects at age<18 years. Diseases affecting the gut microbiota (e.g. chronic diarrhea, Crohn's disease, or ulcerative colitis).

Patients on maintenance dialysis, with diabetes or pregnancy, using antibiotics, probiotics, prebiotics, or synbiotics in the previous 4 weeks.

Patients with critical condition (hypertension emergency,urgency, acute myocardial infarction or stroke within the last 6 months) and suspected/confirmed renal vascular disease.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Female patients at the of child bearing period
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate dysbiosis of some intestinal microbiota in adult patients with lupus nephritis compared to healthy controls. | 2 years
  Evaluate the relation of dysbiosis of some intestinal microbiota to the stage of lupus nephritis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang A, Zhao J, Qin Y, Zhang Y, Xing Y, Wang Y, Yu Z, Yan J, Han M, Yuan J, Hui Y, Guo S, Ning X, Sun S. Alterations of the gut microbiota in the lupus nephritis: a systematic review. Ren Fail. 2023;45(2):2285877. doi: 10.1080/0886022X.2023.2285877. Epub 2023 Nov 23. PMID 37994423